CLINICAL TRIAL: NCT04229017
Title: Safety and Effectiveness of Posterior Cervical Stabilization System (PCSS) as an Adjunct to Posterior Cervical Fusion, When Used in Combination With ACDF in Treatment of Multi-level Cervical Degenerative Disease
Brief Title: Study of Posterior Cervical Stabilization System (PCSS) as Part of Circumferential Fusion to Treat Multilevel DDD
Acronym: FUSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMT0003
Record Dates: First submitted 2019-12-23; First posted 2020-01-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2024-11

CONDITIONS: Degenerative Disc Disease
Keywords: cervical spine; myelopathy; radiculopathy; cervical spine fusion; circumferential cervical fusion; degenerative disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Cord Diseases; Radiculopathy; Klippel-Feil Syndrome | interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled multi-center trial
Who Masked: Participant
Masking Description: Patients will be randomly assigned to either the treatment or control arms at 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anterior Cervical Discectomy and Fusion (ACDF) (Active Comparator): ACDF is a a standard of care procedure that is performed using standard instruments and completed with an allograft interbody implant and anterior plate. The plate is intended to stabilize the treated levels until fusion occurs.
  Interventions: Procedure: Anterior Cervical Discectomy and Fusion
- Circumferential Cervical Fusion (CCF) (Experimental): Circumferential Cervical Fusion (CCF) is a combination of ACDF and Posterior Cervical Fusion (PCF) procedures. The PCF is completed with Posterior Cervical Stabilization System (PCSS).
  Interventions: Device: Posterior Cervical Stabilization System (PCSS)

INTERVENTIONS:
Procedure: Anterior Cervical Discectomy and Fusion — Anterior Cervical Decompression and Fusion (ACDF) is a standard of care procedure that is performed using standard instruments and completed with an allograft interbody implant and anterior plate.
  Other Names: ACDF
  Arms: Anterior Cervical Discectomy and Fusion (ACDF)
Device: Posterior Cervical Stabilization System (PCSS) — Posterior Cervical Stabilization System (PCSS) is non-segmental instrumentation with integrated screw fixation intended to provide immobilization and stabilization of spinal segments. PCSS achieves bilateral facet fixation by spanning the interspace at each level with points of fixation at each end of the construct.
  Arms: Circumferential Cervical Fusion (CCF)

SUMMARY:
This study will evaluate the safety and effectiveness of a device called "Posterior Cervical Stabilization System or PCSS" when used along with posterior cervical fusion (PCF) in combination with anterior cervical discectomy and fusion (ACDF) in the treatment of multi-level cervical degenerative disease.

DETAILED DESCRIPTION:
Degenerative disc disease (DDD) is a condition in which people experience pain because of compression on the spinal cord or nerve roots caused by degenerating cervical discs. Discs sit between the bones of the spine to provide cushioning, shock absorption, mobility, and load-bearing. When the discs break down, the space between the bones gets smaller and squeezes on the spinal cord or nerve roots causing radiating pain down the neck, shoulders, or arms.

A surgical approach to address cervical (neck) DDD is to fuse the bones together to prevent further compression. This can be done with or without removing the disc material itself. The most common way to perform a cervical spinal (neck) fusion to address DDD is to come in from the front of the neck, decompress the spine to relieve pain, and fuse the bones together to prevent further pain in a procedure called Anterior Cervical Discectomy and Fusion (ACDF). Another option is to come in from the back of the neck in a procedure called Posterior Cervical Fusion (PCF). Sometimes these procedures are combined to provide further decompression and stability in the bones of the neck to promote fusion leading to quicker pain relief and return to function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years (Skeletally Mature)
2. Indicated for ACDF treatment of degenerative disc disease (DDD) between and including C3-C7 at 3 contiguous levels
3. NDI Score of ≥15/50
4. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics)
5. Reported to be medically cleared for surgery
6. Physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.
7. Written informed consent provided by subject

Exclusion Criteria:

1. Body Mass Index (BMI) greater than 40 kg/m2
2. Active systemic infection or infection at the operative site
3. History of or anticipated treatment for active systemic infection, including HIV or Hepatitis C
4. Previous trauma to the C3 to C7 levels resulting in significant bony or disco- ligamentous cervical spine injury that may prevent device placements
5. A prior spine surgery or pseudoarthrosis at the operative levels
6. Axial neck pain in the absence of other symptoms of radiculopathy or myeloradiculopathy justifying the need for surgical intervention
7. Symptomatic DDD or significant cervical spondylosis at more than three levels
8. Diagnosis of spondylolisthesis, grade >2
9. Overt (Segmental) instability measured as a movement on dynamic flex/ext x-rays >3.5 mm
10. Congenital bony and/or spinal cord abnormalities that affect spinal stability
11. Diagnosis of Paget's disease, osteomalacia or any other metabolic bone disease other than osteoporosis
12. Osteoporosis, defined as either the SCORE or MORES ≥ 6 and a DEXA bone density measured T-score of ≤ -2.5
13. Active malignancy or a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and without clinical signs or symptoms of the malignancy for at least five years
14. Has an uncontrolled seizure disorder
15. Use of epidural steroids within 14 days prior to surgery
16. A concomitant condition requiring daily, high-dose oral and/or inhaled steroids
17. Known allergy to titanium (Ti).
18. Fixed or permanent neurologic deficit related to the target treatment levels that cannot be improved with surgical decompression
19. Has, in the Investigator's opinion, any disease or condition that would preclude accurate clinical evaluation (e.g. neuromuscular disorders).
20. Is pregnant or nursing at time of screening, or with plans to become pregnant within the next three years.
21. A current or recent history (≤ 1 year prior to screening) of substance abuse (alcoholism and/or narcotic addiction) that required treatment.
22. Long term use (>6 months) of opioids (max. daily amount=120 mg morphine equivalents).
23. A mental illness or belongs to a vulnerable population, as determined by the investigator (e.g., prisoner or developmentally disabled), that would compromise ability to provide informed consent or compliance with follow-up requirements.
24. Any other condition or anatomy (e.g. fused facet) that makes posterior fusion treatment infeasible
25. Use of any other investigational drug or medical device within the last 30 days prior to surgery.
26. A pending personal litigation relating to spinal injury (worker's compensation is not exclusionary).
27. Anticipated or potential relocation greater than 50 miles that may interfere with completion of follow-up examinations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Superiority in Fusion Success in CCF (treatment) compared to ACDF (control) | 12 months
  An individual subject is considered a fusion success if there is evidence of bridging trabecular bone across endplates and < 2° total angular motion

SECONDARY OUTCOMES:
Non-inferiority Composite Safety Success in CCF (treatment) compared to ACDF (control) | 24 months
  An individual subject is considered a success if all of the following safety criteria are met:
  1. Fusion success - as defined by evidence of bridging trabecular bone across endplates and < 2° total angular motion
  2. Improvement in Neck Disability Index (NDI)
  3. Improvement in Neurological function
  4. Absence of secondary surgical interventions (SSI)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Jenkins, Study Director — Providence Medical Technology, Inc.
Locations (17):
- United States (17):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Scripps, Encinitas, California
  - OrthoNorCal, Los Gatos, California
  - Spine Colorado, Durango, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - The Orthopaedic Institute, Paducah, Kentucky
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - LSU Health, New Orleans, Louisiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - LifeBridge Health - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Beaumont Health, Royal Oak, Michigan
  - Inspira Health Network, Vineland, New Jersey
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - Atlantic Neurosurgical & Spine Specialists, Wilmington, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas